CLINICAL TRIAL: NCT01082549
Title: Randomized Phase 3 Trial of Gemcitabine/Carboplatin With or Without Iniparib (SAR240550) (a PARP1 Inhibitor) in Subjects With Previously Untreated Stage IV Squamous Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Trial of Gemcitabine/Carboplatin With or Without Iniparib (SAR240550) (a PARP1 Inhibitor) in Subjects With Previously Untreated Stage IV Squamous Non-Small-Cell Lung Cancer (NSCLC)
Acronym: ECLIPSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11553; 20090321 (Other: Bipar code)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Patients with Previously Untreated Advanced Squamous Cell Lung Cancer
MeSH Terms: interventions — Gemcitabine; Carboplatin; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine/carboplatin (Active Comparator)
  Interventions: Drug: gemcitabine/carboplatin
- gemcitabine/carboplatin plus Iniparib (Experimental)
  Interventions: Drug: gemcitabine/carboplatin plus Iniparib

INTERVENTIONS:
Drug: gemcitabine/carboplatin — i.v.
  Arms: gemcitabine/carboplatin
Drug: gemcitabine/carboplatin plus Iniparib — i.v.
  Arms: gemcitabine/carboplatin plus Iniparib

SUMMARY:
To evaluate the overall survival (OS) of patients with advanced squamous cell lung cancer receiving the combination of gemcitabine/carboplatin either with or without Iniparib.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must meet the following criteria to be enrolled in the study:

1. Newly diagnosed, stage IV squamous cell lung cancer. This includes patients who present with disseminated metastases, and those with a malignant pleural or pericardial effusion (i.e., formerly stage IIIB in the 6th TNM staging system).
2. Patients who have received prior adjuvant therapy for early-stage lung cancer are eligible if at least 12 months have elapsed from that treatment.
3. Histologically confirmed squamous cell bronchogenic carcinoma. Patients whose tumors contain mixed non-small cell histologies are eligible, as long as squamous carcinoma is the predominant histology. Mixed tumors with small cell anaplastic elements are not eligible. Cytologic specimens obtained by brushings, washings, or needle aspiration of the defined lesion are acceptable.
4. Patients with previous radiotherapy as definitive therapy for locally advanced non-small cell lung cancer are eligible, as long as the recurrence is outside the original radiation therapy port. Radiation therapy must have been completed >4 weeks prior to the initiation of study treatment. Patients who have received chemo/radiation for locally advanced NSCLC are not eligible. Patients who have received palliative radiation therapy for symptomatic metastases must have completed treatment >14 days prior the initiation of the study treatment.
5. Presence of evaluable (measureable or non-measurable) disease.
6. ECOG Performance Status of 0 or 1.
7. Laboratory values as follows:

   * Absolute neutrophil count (ANC) >1,500/microL and platelets >100,000/microL (≤72 hours prior to initial treatment).
   * Hemoglobin >9 g/dL (Note: Patients may be transfused or receive erythropoietin to maintain or exceed this level).
   * Bilirubin < ULN.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal if no liver involvement or ≤5 times the upper limit of normal with liver involvement.
   * Creatinine <2.0 mg/dL, or creatinine clearance >40 mL/min (as calculated by the Cockcroft-Gault method.
8. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment and at least 6 months after the last dose of the study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately. Sexually active men must agree to use a medically acceptable form of birth control during treatment and at least 6 months after the last dose. If a female partner becomes pregnant during the course of the study the treating physician should be informed immediately.
9. >18 years of age.
10. Ability to understand the nature of this study, give written informed consent, and comply with study requirements.
11. Patients entering this study must be willing to provide tissue from a previous tumor biopsy (if available) for correlative testing. An exception to this is when the national/local regulations prohibits some of the key activities of this research like the export of samples to third countries, storage of coded samples or global gene expression profiling without a pre-specified list of target genes. If tissue is not available, a patient will still be eligible for enrollment into the study.

Exclusion Criteria:

1. Prior treatment with gemcitabine, carboplatin (except in the adjuvant setting), or Iniparib.
2. Past or current history of neoplasm other than the entry diagnosis, with the exception of treated non-melanoma skin cancer or carcinoma in-situ of any primary site, or invasive cancers treated definitively, with treatment ending >5 years previously and no evidence of recurrences.
3. A history of cardiac disease, as defined by:

   * Malignant hypertension
   * Unstable angina
   * Congestive heart failure
   * Myocardial infarction within the previous 6 months
   * Symptomatic, unstable or uncontrolled, cardiac arrhythmias. Patients who have stable, rate-controlled atrial fibrillation are eligible for study enrollment.
4. Active brain metastases. Patients with treated brain metastases are eligible, if (1) radiation therapy was completed at least 2 weeks prior to study entry; (2) follow-up scan shows no disease progression; and (3) patient does not require steroids.
5. Women who are pregnant or lactating.
6. Any serious, active infection (> Grade 2) at the time of treatment.
7. A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
8. A major surgical procedure, or significant traumatic injury ≤28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study.
9. Uncontrolled or intercurrent illness including, that in the opinion of the investigator may increase the risks associated with study participation or administration of the investigational products, or that may interfere with the interpretation of the results.
10. History of any medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with the study participation or administration of the investigational products, or that may interfere with the interpretation of the results.
11. Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
overall survival | 12 months, 24 months

SECONDARY OUTCOMES:
progression free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (142):
- United States (67):
  - Investigational Site Number 840306, Birmingham, Alabama
  - Investigational Site Number 840207, Huntsville, Alabama
  - Investigational Site Number 840351, Muscle Shoals, Alabama
  - Investigational Site Number 840338, Anaheim, California
  - Investigational Site Number 840353, Burbank, California
  - Investigational Site Number 840341, Concord, California
  - Investigational Site Number 840317, Duarte, California
  - Investigational Site Number 840339, La Verne, California
  - Investigational Site Number 840309, Loma Linda, California
  - Investigational Site Number 840307, Los Angeles, California
  - Investigational Site Number 840327, Maywood, California
  - Investigational Site Number 840303, San Diego, California
  - Investigational Site Number 840321, Santa Rosa, California
  - Investigational Site Number 840326, Stockton, California
  - Investigational Site Number 840310, Vallejo, California
  - Investigational Site Number 840336, Denver, Colorado
  - Investigational Site Number 840346, Norwich, Connecticut
  - Investigational Site Number 840315, Newark, Delaware
  - Investigational Site Number 840216, Fort Lauderdale, Florida
  - Investigational Site Number 840215, Jacksonville, Florida
  - Investigational Site Number 840217, Lakeland, Florida
  - Investigational Site Number 840205, Orlando, Florida
  - Investigational Site Number 840104, Sarasota, Florida
  - Investigational Site Number 840343, Athens, Georgia
  - Investigational Site Number 840213, Augusta, Georgia
  - Investigational Site Number 840347, Augusta, Georgia
  - Investigational Site Number 840201, Gainesville, Georgia
  - Investigational Site Number 840301, Lawrenceville, Georgia
  - Investigational Site Number 840305, Marietta, Georgia
  - Investigational Site Number 840314, Tucker, Georgia
  - Investigational Site Number 840313, Chicago, Illinois
  - Investigational Site Number 840218, Evansville, Indiana
  - Investigational Site Number 840319, Indianapolis, Indiana
  - Investigational Site Number 840329, South Bend, Indiana
  - Investigational Site Number 840316, Wichita, Kansas
  - Investigational Site Number 840320, Louisville, Kentucky
  - Investigational Site Number 840308, Scarborough, Maine
  - Investigational Site Number 840202, Bethesda, Maryland
  - Investigational Site Number 840345, Salisbury, Maryland
  - Investigational Site Number 840337, Royal Oak, Michigan
  - Investigational Site Number 840328, Saint Louis Park, Minnesota
  - Investigational Site Number 840210, Bridgeton, Missouri
  - Investigational Site Number 840212, Omaha, Nebraska
  - Investigational Site Number 840318, Las Vegas, Nevada
  - Investigational Site Number 840204, Morristown, New Jersey
  - Investigational Site Number 840350, Chapel Hill, North Carolina
  - Investigational Site Number 840330, Durham, North Carolina
  - Investigational Site Number 840105, Cincinnati, Ohio
  - Investigational Site Number 840302, Cleveland, Ohio
  - Investigational Site Number 840348, Cleveland, Ohio
  - Investigational Site Number 840335, Columbus, Ohio
  - Investigational Site Number 840311, Bend, Oregon
  - Investigational Site Number 840211, West Reading, Pennsylvania
  - Investigational Site Number 840352, Charleston, South Carolina
  - Investigational Site Number 840106, Columbia, South Carolina
  - Investigational Site Number 840220, Spartanburg, South Carolina
  - Investigational Site Number 840103, Chattanooga, Tennessee
  - Investigational Site Number 840208, Chattanooga, Tennessee
  - Investigational Site Number 840203, Collierville, Tennessee
  - Investigational Site Number 840101, Nashville, Tennessee
  - Investigational Site Number 840323, Fort Worth, Texas
  - Investigational Site Number 840219, Newport News, Virginia
  - Investigational Site Number 840102, Richmond, Virginia
  - Investigational Site Number 840312, Seattle, Washington
  - Investigational Site Number 840344, Tacoma, Washington
  - Investigational Site Number 840322, Morgantown, West Virginia
  - Investigational Site Number 840331, Wauwatosa, Wisconsin
- Belgium (3):
  - Investigational Site Number 056004, Bruges
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056001, Liège
- Canada (6):
  - Investigational Site Number 124003, Edmonton
  - Investigational Site Number 124006, Greenfield Park
  - Investigational Site Number 124005, London
  - Investigational Site Number 124007, Oshawa
  - Investigational Site Number 124004, Québec
  - Investigational Site Number 124001, Toronto
- France (10):
  - Investigational Site Number 250007, Brest
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250009, Limoges
  - Investigational Site Number 250003, Marseille
  - Investigational Site Number 250004, Paris
  - Investigational Site Number 250010, Pierre-Bénite
  - Investigational Site Number 250008, Poitiers
  - Investigational Site Number 250001, Saint-Herblain
  - Investigational Site Number 250006, Strasbourg
  - Investigational Site Number 250005, Tours
- Germany (10):
  - Investigational Site Number 276002, Amberg
  - Investigational Site Number 276004, Berlin
  - Investigational Site Number 276007, Frankfurt am Main
  - Investigational Site Number 276008, Großhansdorf
  - Investigational Site Number 276010, Halle
  - Investigational Site Number 276012, Heidelberg
  - Investigational Site Number 276009, Immenhausen
  - Investigational Site Number 276001, Löwenstein
  - Investigational Site Number 276006, München
  - Investigational Site Number 276003, Oldenburg
- Hungary (4):
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348003, Budapest
  - Investigational Site Number 348001, Mátraháza
  - Investigational Site Number 348004, Nyíregyháza
- Israel (4):
  - Investigational Site Number 376002, Kfar Saba
  - Investigational Site Number 376005, Petah Tikva
  - Investigational Site Number 376003, Tel Litwinsky
  - Investigational Site Number 376001, Tzrifin
- Italy (6):
  - Investigational Site Number 380006, Genova
  - Investigational Site Number 380001, Novara
  - Investigational Site Number 380008, Orbassano
  - Investigational Site Number 380002, Perugia
  - Investigational Site Number 380003, Roma
  - Investigational Site Number 380007, Roma
- Investigational Site Number 442001, Luxembourg, Luxembourg
- Netherlands (5):
  - Investigational Site Number 528005, Breda
  - Investigational Site Number 528004, Eindhoven
  - Investigational Site Number 528001, Groningen
  - Investigational Site Number 528006, Maastricht
  - Investigational Site Number 528003, Zwolle
- Poland (7):
  - Investigational Site Number 616006, Bialystok
  - Investigational Site Number 616001, Krakow
  - Investigational Site Number 616007, Lubin
  - Investigational Site Number 616004, Olsztyn
  - Investigational Site Number 616008, Torun
  - Investigational Site Number 616002, Warsaw
  - Investigational Site Number 616005, Wroclaw
- Romania (5):
  - Investigational Site Number 642002, Alba Iulia
  - Investigational Site Number 642006, Bucharest
  - Investigational Site Number 642001, Cluj-Napoca
  - Investigational Site Number 642004, Craiova
  - Investigational Site Number 642005, Hunedoara
- Spain (10):
  - Investigational Site Number 724004, A Coruña
  - Investigational Site Number 724009, Badalona
  - Investigational Site Number 724003, Barcelona
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724006, Madrid
  - Investigational Site Number 724002, Málaga
  - Investigational Site Number 724001, Palma de Mallorca
  - Investigational Site Number 724008, Seville
  - Investigational Site Number 724010, Valencia
  - Investigational Site Number 724007, Zaragoza
- United Kingdom (4):
  - Investigational Site Number 826002, Glasgow
  - Investigational Site Number 826005, Leeds
  - Investigational Site Number 826001, Manchester
  - Investigational Site Number 826006, Wolverhampton